CLINICAL TRIAL: NCT02810899
Title: The Effect of Dexmedetomidine as an Adjuvant to General Anesthesia on Intelligence Development in Pediatric Patients Undergoing Craniotomy: a Randomized, Double-blind and Placebo-controlled Pilot Trial
Brief Title: Dexmedetomidine and Intelligence Development in Pediatric Patients Undergoing Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015[969]; ChiCTR-IPR-15007085 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2016-06-08; First posted 2016-06-23 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Brain Neoplasms
Keywords: child; craniotomy; intelligence tests; dexmedetomidine; Disruption; Dehiscence; Mild Cognitive Disorder
MeSH Terms: conditions — Brain Neoplasms; Neurocognitive Disorders | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Experimental): A loading dose of dexmedetomidine (0.5 ug/kg IV infusion in 15 minutes) will be administered after induction of general anesthesia, followed by continuous infusion at a rate of 0.5 ug/kg/h until the closure of the duramater of the brain.
  Interventions: Drug: dexmedetomidine
- Control group (Placebo Comparator): Normal saline will be administered in the same rate and volume as that in the dexmedetomidine group.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: dexmedetomidine — A loading dose dexmedetomidine (0.5 ug/kg IV infused in 15 minutes) will be administered after anesthesia induction, followed by a continuous infusion at a rate of 0.5 ug/kg/h until the closure of the brain duramater at the end of surgery.
  Other Names: dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: normal saline — Normal saline will be administered in the same rate, volume and duration as that in the dexmedetomidine group
  Other Names: 0.9% sodium chloride
  Arms: Control group

SUMMARY:
The purpose of this randomized, double-blind and placebo-controlled pilot study is to investigate whether dexmedetomidine when used as an adjuvant to general anesthesia can decrease the harmful effects of anesthesia and surgery on intelligence development in pediatric patients undergoing craniotomy.

DETAILED DESCRIPTION:
General anesthetics and sedatives are administered to millions of children each year to facilitate life-saving surgery and other essential surgical or medical procedures. In the past two decades, mounting evidence from animal and clinical studies have raised concerns that general anesthetics may produce harmful effects in the developing brain and lead to adverse neurodevelopmental outcomes. Factors that may influence the degree of injury include age at the time of drug exposure/surgery and cumulative anesthetic dose.

The Intelligence Quotients of pediatric patients with intracranial tumors are lower when compared with healthy children of same age. The investigators suppose that these patients are more sensitive to the neurotoxic effects of general anesthetics. Dexmedetomidine is an alpha 2-adrenoceptor agonist that provides sedation, anxiolysis, and analgesia, and has been shown to be safe to the brain in animal studies. In clinical studies, the use of dexmedetomidine decreases the consumption of anesthetics and opioids during general anesthesia and suppresses stress response induced by surgery. The investigators hypothesize that dexmedetomidine, when used as an adjuvant to general anesthesia, can reduce the neurotoxic effects of general anesthetics by decreasing anesthetic consumption and inhibiting stress response.

The purpose of this randomized, double-blind and placebo-controlled pilot study is to investigate whether dexmedetomidine, when used as an adjuvant to general anesthesia, can decrease the harmful effects of anesthesia and surgery on intelligence development of pediatric patients undergoing craniotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 2 years or older, but no more than 12 years;
2. Plan to undergo selective craniotomy under general anesthesia for intracranial tumor resection;
3. Written informed consent signed by legal guardians.

Exclusion Criteria:

1. Refused to participate by the legal guardians;
2. Body weight lower than the 3rd percentile or higher than 97th percentile of the normal body weight reference;
3. American Society of Anesthesiologists physical classification of IV or higher;
4. Unable to complete preoperative intelligence assessment because of coma, dysnoesia, or language barrier;
5. Diagnosed pulmonary disease (including acute respiratory tract infection) or cardiovascular disease (including congenital heart disease, hypertension, hypotension, bradycardia, atrioventricular block, or cardiac insufficiency);
6. Abnormal liver or renal function (liver enzyme or creatinine higher than 1.5 times of the upper normal limit;
7. Other congenital diseases that may affect the development of the nervous system (such as Down's Syndrome);
8. Allergy to dexmedetomidine;
9. Other conditions that are considered unsuitable for study participation by the attending pediatricians or investigators.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Intelligence Quotient | At 3 months after surgery
  Tested with Chinese Binet Intelligence Scale

SECONDARY OUTCOMES:
Time to anesthesia emergence | From end of surgery until reappearance of response to oral orders, assessed up to 24 hours
Time to extubation | From end of surgery until extubation, assessed up to 24 hours
Depth of sedation at the time of extubation | Immediately after extubation
  Assessed with Ramsay sedation scale
Emergence agitation | From end of surgery until extubation, assessed up to 24 hours
  Agitation will be assessed with anesthesia emergence agitation score.

OTHER OUTCOMES:
Length of stay in hospital after surgery | From end of surgery to 30 days after surgery
Incidence of postoperative complications | From end of surgery to 30 days after surgery
All-cause 30-day mortality | At the time of 30 days after surgery
All-cause 90-day mortality | At the time of 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rappaport BA, Suresh S, Hertz S, Evers AS, Orser BA. Anesthetic neurotoxicity--clinical implications of animal models. N Engl J Med. 2015 Feb 26;372(9):796-7. doi: 10.1056/NEJMp1414786. PMID 25714157
- [Background] Cattano D, Young C, Straiko MM, Olney JW. Subanesthetic doses of propofol induce neuroapoptosis in the infant mouse brain. Anesth Analg. 2008 Jun;106(6):1712-4. doi: 10.1213/ane.0b013e318172ba0a. PMID 18499599
- [Background] Ikonomidou C, Bosch F, Miksa M, Bittigau P, Vockler J, Dikranian K, Tenkova TI, Stefovska V, Turski L, Olney JW. Blockade of NMDA receptors and apoptotic neurodegeneration in the developing brain. Science. 1999 Jan 1;283(5398):70-4. doi: 10.1126/science.283.5398.70. PMID 9872743
- [Background] Olney JW, Ishimaru MJ, Bittigau P, Ikonomidou C. Ethanol-induced apoptotic neurodegeneration in the developing brain. Apoptosis. 2000 Dec;5(6):515-21. doi: 10.1023/a:1009685428847. PMID 11303910
- [Background] Jevtovic-Todorovic V, Absalom AR, Blomgren K, Brambrink A, Crosby G, Culley DJ, Fiskum G, Giffard RG, Herold KF, Loepke AW, Ma D, Orser BA, Planel E, Slikker W Jr, Soriano SG, Stratmann G, Vutskits L, Xie Z, Hemmings HC Jr. Anaesthetic neurotoxicity and neuroplasticity: an expert group report and statement based on the BJA Salzburg Seminar. Br J Anaesth. 2013 Aug;111(2):143-51. doi: 10.1093/bja/aet177. Epub 2013 May 30. PMID 23722106
- [Background] Poggi G, Liscio M, Galbiati S, Adduci A, Massimino M, Gandola L, Spreafico F, Clerici CA, Fossati-Bellani F, Sommovigo M, Castelli E. Brain tumors in children and adolescents: cognitive and psychological disorders at different ages. Psychooncology. 2005 May;14(5):386-95. doi: 10.1002/pon.855. PMID 15386759
- [Background] Hernandez MT, Sauerwein HC, Jambaque I, de Guise E, Lussier F, Lortie A, Dulac O, Lassonde M. Attention, memory, and behavioral adjustment in children with frontal lobe epilepsy. Epilepsy Behav. 2003 Oct;4(5):522-36. doi: 10.1016/j.yebeh.2003.07.014. PMID 14527495
- [Background] Wang XW, Cao JB, Lv BS, Mi WD, Wang ZQ, Zhang C, Wang HL, Xu Z. Effect of perioperative dexmedetomidine on the endocrine modulators of stress response: a meta-analysis. Clin Exp Pharmacol Physiol. 2015 Aug;42(8):828-36. doi: 10.1111/1440-1681.12431. PMID 26016707
- [Background] Li Y, Wang B, Zhang LL, He SF, Hu XW, Wong GT, Zhang Y. Dexmedetomidine Combined with General Anesthesia Provides Similar Intraoperative Stress Response Reduction When Compared with a Combined General and Epidural Anesthetic Technique. Anesth Analg. 2016 Apr;122(4):1202-10. doi: 10.1213/ANE.0000000000001165. PMID 26991622
- [Background] Kim DJ, Kim SH, So KY, Jung KT. Effects of dexmedetomidine on smooth emergence from anaesthesia in elderly patients undergoing orthopaedic surgery. BMC Anesthesiol. 2015 Oct 7;15:139. doi: 10.1186/s12871-015-0127-4. PMID 26446479
- [Background] Le Bot A, Michelet D, Hilly J, Maesani M, Dilly MP, Brasher C, Mantz J, Dahmani S. Efficacy of intraoperative dexmedetomidine compared with placebo for surgery in adults: a meta-analysis of published studies. Minerva Anestesiol. 2015 Oct;81(10):1105-17. Epub 2015 May 25. PMID 26005187